CLINICAL TRIAL: NCT04972396
Title: An Open-label Study of the Effect of ALT-801 on the Pharmacokinetics of Metformin, Warfarin, Atorvastatin, Digoxin, and the Combined Oral Contraceptive Ethinylestradiol/Levonorgestrel in Healthy Volunteers
Brief Title: Pemvidutide (ALT-801) DDI Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ALT-801-103; Pemvidutide (Other: Altimmune); ALT-801 (Other: Altimmune)
Record Dates: First submitted 2021-07-14; First posted 2021-07-22 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — ALT-801; Metformin; Atorvastatin; Warfarin; Digoxin; Ethinyl Estradiol; Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part 1 Metformin and Atorvastatin with and without Pemvidutide (Experimental): In Period 1, subjects received metformin 500 mg BID on Days 1 and 2, single doses of metformin 500 mg and atorvastatin 40 mg on Day 3, and a single dose of pemvidutide 0.6 mg on Day 8.
  In Period 2, subjects received single doses of pemvidutide1.2 mg on Day 15 and 1.8 mg on Days 22 and 29, metformin 500 mg BID on Days 34 and 35, and pemvidutide 1.8 mg on Day 36 immediately followed by oral metformin 500 mg and atorvastatin 40 mg.
  Interventions: Drug: Pemvidutide; Drug: Metformin; Drug: Atorvastatin
- Part 2 Warfarin and Digoxin with and without Pemvidutide (Experimental): In Period 1, subjects received single doses of warfarin 10 mg and digoxin 500 mcg (0.5 mg) on Day 1, and a single dose of pemvidutide 0.6 mg on Day 8.
  In Period 2, subjects received single doses of pemvidutide 1.2 mg on Day 15 and 1.8 mg on Days 22 and 29, and pemvidutide1.8 mg immediately followed by warfarin 10 mg and digoxin 500 mcg (0.5 mg) on Day 36.
  Interventions: Drug: Pemvidutide; Drug: Warfarin; Drug: Digoxin
- Part 3 Ethinylestradiol and Levonorgestrel with and without Pemvidutide (Experimental): In Period 1, subjects received a combined oral contraceptive (COC) consisting of 0.03 mg ethinylestradiol and 0.15 mg levonorgestrel once daily on Days 1 through 9 and a single dose of pemvidutide 0.6 mg on Day 15.
  In Period 2, subjects received single doses of pemvidutide 1.2 mg on Day 22 and 1.8 mg on Days 29 and 36. Subjects also received COC once daily on Days 35 through 42 and a single dose of pemvidutide 1.8 mg followed immediately by a single dose of COC on Day 43.
  Interventions: Drug: Pemvidutide; Drug: Ethinylestradiol and Levonorgestrel

INTERVENTIONS:
Drug: Pemvidutide — Injected subcutaneously (SC)
  Other Names: ALT-801
Drug: Metformin — Taken by mouth (PO)
  Arms: Part 1 Metformin and Atorvastatin with and without Pemvidutide
Drug: Atorvastatin — Taken by mouth (PO)
  Arms: Part 1 Metformin and Atorvastatin with and without Pemvidutide
Drug: Warfarin — Taken by mouth (PO)
  Arms: Part 2 Warfarin and Digoxin with and without Pemvidutide
Drug: Digoxin — Taken by mouth (PO)
  Arms: Part 2 Warfarin and Digoxin with and without Pemvidutide
Drug: Ethinylestradiol and Levonorgestrel — Taken by mouth (PO)
  Arms: Part 3 Ethinylestradiol and Levonorgestrel with and without Pemvidutide

SUMMARY:
This is a Phase 1, open-label, drug-drug interaction (DDI) study of pemvidutide (ALT-801) under steady state conditions on concomitantly administered medications in healthy subjects. The study will evaluate the effect of pemvidutide on the pharmacokinetics (PK) of metformin, warfarin, atorvastatin, digoxin, and the combined oral contraceptive (COC) ethinylestradiol/levonorgestrel. The study will be conducted in 3 parts, as described below. Each part will have 2 periods in a fixed sequence, where the first period is without pemvidutide administration and the second is with pemvidutide at steady state.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy volunteers, age 18 to 55 years, inclusive
* Body mass index (BMI) 28.0- 40.0 kg/m2
* Able and willing to provide written informed consent prior to entry into the study

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* History of diabetes or use of medications for the treatment of diabetes, or hyperglycemia or HbA1c ≥ 6.5%
* History of pancreatitis or hypersensitivity reaction to GLP-1 analogues

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) of metformin and atorvastatin/warfarin and digoxin in presence of steady state ALT-801 | Baseline and Day 36
Area Under the Plasma Concentration Versus Time Curve (AUC) of ethinylestradiol and levonorgestrel in presence of steady state ALT-801 | Baseline and Day 43

SECONDARY OUTCOMES:
Cmax and Tmax of metformin and atorvastatin/warfarin and digoxin | Day 36
Cmax and Tmax of ethinylestradiol and levonorgestrel | Day 43
The Number of Participants with One or More Treatment-Emergent Adverse Events (TEAEs) | Up to Day 77

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - CMAX Clinical Research, Adelaide, South Australia
  - Nucleus Network, Brisbane